CLINICAL TRIAL: NCT00158184
Title: Prescription Opioid Effects in Drug and Non-drug Abusers - 1
Brief Title: Prescription Opioid Effects in Abusers Versus Non-Abusers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: #4691; R01DA016759-01 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: Opiate; Opioid; Abuse Liability; Abuse Potential
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rx Opioid Abusers (Active Comparator): Recreational users of prescription opioids. Participants in this arm received the 3 interventions (0, 15, and 30 mg oxycodone) at random.
  Interventions: Drug: oxycodone 15 mg; Drug: oxycodone 30 mg; Drug: Placebo 0 mg
- Rx Opioid Non-Abusers (Active Comparator): Participants with a history of prescription opioid use, but who did not abuse them. Participants in this arm received the 3 interventions (0, 15, and 30 mg) at random.
  Interventions: Drug: oxycodone 15 mg; Drug: oxycodone 30 mg; Drug: Placebo 0 mg

INTERVENTIONS:
Drug: oxycodone 15 mg — 15 mg/70 kg oxycodone administered once per day, orally.
  Other Names: immediate-release oxycodone
Drug: oxycodone 30 mg — 30 mg/70 kg oxycodone administered once per day, orally.
  Other Names: immediate-release oxycodone
Drug: Placebo 0 mg — 0 mg placebo dose administered once a day, orally.
  Other Names: 0 mg

SUMMARY:
The purpose of this study is to examine the abuse liability of oxycodone in individuals with, and without, a history of prescription opioid abuse.

DETAILED DESCRIPTION:
Prescription opioid abuse is becoming an increasingly widespread and serious public health concern. The 2001 National Household Survey on Drug Abuse report revealed that the number of first-time users of prescription opioid medications for non-medical reasons reached 2 million in the year 2000, a number that has quintupled since 1984. Despite this trend, little experimental research has been directed towards understanding who may be abusing these medications, and under what conditions. The study will examine the reinforcing, subjective, performance, and physiological effects of oxycodone. Because it is not clear who is abusing prescription opioids, the medication effects will be compared in drug abusers and non-drug abusers.

ELIGIBILITY:
Inclusion Criteria:

* In good physical health
* Women reporting regular menstrual cycles lasting between 24 to 35 days
* Able to perform study procedures
* Normal body weight
* Use of opioids for medical purposes (cough, pain, or diarrhea) or recreational purposes at least twice in lifetime with no serious adverse effects
* Current opioid abuse, but not opioid dependence (drug abusers only)

Exclusion Criteria:

* On parole or probation
* Recently convicted of a crime of violence
* History of significant violent behavior
* Current Axis I psychopathology
* Significant Axis II disorder
* Pregnancy
* Women who have irregular menstrual cycles, or who are dysmenorrheic, amenorrheic, or menopausal
* Women who have been pregnant or breastfeeding within the past 6 months
* Women who have had a miscarriage or abortion within the past 6 months
* Women who meet DSM-IV criteria for premenstrual dysphoric disorder
* Women who report suffering from moderate to severe premenstrual symptoms
* Women seeking treatment for premenstrual problems
* Taking prescription or over-the-counter psychotropic medication
* History of chronic pain, or routinely uses over-the-counter analgesics (more than 4 days per month)
* Blood pressure greater than 150/90 mm Hg
* Reports of sensitivity, allergy, or contraindication to opioids
* Non-drug abusers:

  1. Current or lifetime history of substance abuse or dependence according to DSM-IV criteria (those requiring detoxification)
  2. Consumes more than 500 mg caffeine daily
  3. Seeking treatment for substance use

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Comer, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Comer SD, Sullivan MA, Vosburg SK, Kowalczyk WJ, Houser J. Abuse liability of oxycodone as a function of pain and drug use history. Drug Alcohol Depend. 2010 Jun 1;109(1-3):130-8. doi: 10.1016/j.drugalcdep.2009.12.018. Epub 2010 Jan 15. PMID 20079977

RESULTS

PARTICIPANT FLOW:
Groups:
- Rx Opioid Abusers: The Abuse potential 3 doses of oral oxycodone (0, 15, 30 mg) were tested among a group of recreational prescription opioid (Rx) users.
- Rx Opioid Non-Abusers: The Abuse potential 3 doses of oral oxycodone (0, 15, 30 mg) were tested among a group of participants with no history of opioid abuse.
Period: Overall Study
Arm/Group | Rx Opioid Abusers | Rx Opioid Non-Abusers
Started | 16 | 11
Completed | 10 | 9
Not Completed | 6 | 2
Not completed — personal issues | 3 | 1
Not completed — failed for follow unit/study rules | 2 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Rx Opioid Abusers: Prescription Opioids users with abusive patterns of use.
- Rx Opioid Medical Users: Prescription Opioids users without abusive patterns of use.
- Total: Total of all reporting groups
Arm/Group | Rx Opioid Abusers | Rx Opioid Medical Users | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8) | 28 (6) | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Breakpoint
Description: Maximum number of finger presses on a computer mouse completed. The "Breakpoint" is the amount of work (clicks on a mouse) participants were willing to do in order to received the dose of drug under investigation. This is a commonly used indicator of a drugs value and abuse liability.
Time Frame: Measured at 0, 60, 120, 180 and 240 minutes following administration of each oral oxycodone dose (0 , 15, 30 mg). Results presented as mean of the session
Measure: Mean (Standard Error); unit: Mouse Clicks
Groups:
- Rx Opioid Abusers: Recreational prescription opioid users.
- Rx Opioid Non-Abusers: Medical prescription opioid users.
Arm/Group | Rx Opioid Abusers | Rx Opioid Non-Abusers
Number analyzed (Participants) | 10 | 9
Mouse Clicks
  Placebo: 0 mg | 25 (20) | 400 (200)
  Oxycodone: 15mg | 1400 (400) | 850 (100)
  Oxycodone: 30mg | 1100 (350) | 900 (160)

2. Secondary Outcome: Drug Liking
Description: Subjective rating of drug "Liking" on a scale of 0 to 100. Greater numbers indicate greater subjective report of "Liking."
Time Frame: Highest rating obtained following adminstration of each of the 3 test doses.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Rx Opioid Abusers: Recreation users
- Rx Opioid Non-Abusers: Medical users
Arm/Group | Rx Opioid Abusers | Rx Opioid Non-Abusers
Number analyzed (Participants) | 10 | 9
units on a scale
  Placebo: 0 mg | 23 (5) | 21 (7)
  Oxycodone: 15 mg | 60 (7) | 53 (8)
  Oxycodone: 30 mg | 59 (8) | 40 (9)

ADVERSE EVENTS:
Time Frame: Averse events were assessed daily from the date of admission until the date of discharge. Participants also returned for a 30-Day follow-up after being discharged, during which adverse events were assessed.
Description: Adverse events are classified as serious or non-serious.
Arm/Group | Rx Opioid Abusers | Rx Opioid Non-Abusers
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 2/16 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rx Opioid Abusers (N=16) | Rx Opioid Non-Abusers (N=11)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Occurred after admission but prior to oral oxycodone being given.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No